CLINICAL TRIAL: NCT03332407
Title: Does Preoperative Sleep Quality Affect the Postoperative Emergence Delirium in Children Undergoing Strabismus Surgery?
Brief Title: Does Preoperative Sleep Quality Affect the Postoperative Emergence Delirium in Children Undergoing Strabismus Surgery
Status: Completed | Type: Observational
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeon-Jeong Lee, Associated professor, Pusan National University Hospital
Other Study IDs: 2017-1022
Record Dates: First submitted 2017-10-22; First posted 2017-11-06 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Delirium; Strabismus; Sleep Disorder
Keywords: Postoperative delirium; Sleep quality; Pediatric anesthesia; Strabismus surgery
MeSH Terms: conditions — Emergence Delirium; Strabismus; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep is important in maintaining the physiological function of the human body. Recently several studies have reported that preoperative sleep quality is associated with postoperative emergence delirium (ED) The ED is a common in pediatric patients undergoing general anesthesia with sevoflurane, but studies on the association of sleep quality have been rare. The investigators, therefore, aimed to investigate the relationship between postoperative delirium and pre and postoperative sleep quality in pediatric patients receiving strabismus surgery through this study

DETAILED DESCRIPTION:
This study aimed on pediatric patients aged 4-12 years, undergoing elective strabismus surgery. Informed consent was obtained from both parents and children on the day of pre-anesthetic evaluation visit. The child and his or her parents were questioned on preoperative patient's sleep quality based on Pittsburg Sleep Quality Index (PSQI). Surgery was performed under the same anesthesia as usual. After the operation, extubation was performed and patient was moved to post anesthesia recovery room (PACU). During the stay in PACU, one investigator measured degree of ED by Watcha and PAED (Post anesthesia emergence delirium ) scale to minimize bias. One day after the surgery, the investigator mede a phone call to the parents of the patient to obtain information for postoperative PSQI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children without any underlying diseases
* 4~12 years old
* Undergoing strabismus surgery

Exclusion Criteria:

* Any underlying diseases
* Disagree

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subject of this study is pediatric patients aged 4~12 years, undergoing elective strabismus surgery.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Preoperative Pittsburgh Sleep Quality Index(PSQI) | 1. Before the surgery ( Within a week before the surgery)
  1. Add the Seven component score. Score range : 0~27
  2. A total score of "5" or greater is indicative of poor sleep quality.
Watcha scale (For emergence delirium) | 20 min after awakening ( In the post anesthesia recovery room)
  1. Measure the score of most appropriate state of condition. There are four conditions. Score range : 1~4
  2. The score of "3" or greater is indicative of emergence delirium
Pediatric anesthesia emergence delirium scale (PAED) scale | 20 min after awakening ( In the post anesthesia recovery room)
  1. Add the five component score. Score range : 0~20
  2. A total score of "10" or greater is indicative of emergence delirium.
Postoperative Pittsburgh Sleep Quality Index(PSQI) | 1 day after the surgery ( < 24 hours )
  1. Add the Seven component score. Score range : 0~27
  2. A total score of "5" or greater is indicative of poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan national university hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Do W, Kim HS, Kim SH, Kang H, Lee D, Baik J, Lee HJ, Hong JM. Sleep quality and emergence delirium in children undergoing strabismus surgery: a comparison between preschool- and school-age patients. BMC Anesthesiol. 2021 Nov 22;21(1):290. doi: 10.1186/s12871-021-01507-2. PMID 34809579